CLINICAL TRIAL: NCT00511979
Title: Effect of Different Doses of Inhaled Technosphere Insulin on Glucose Infusion Rates During Euglycemic Clamps in Comparison to a Subcutaneous Injection of Regular Human Insulin
Brief Title: Comparison of the Effect on the Glucose Infusion Rates Between Inhaled Technosphere Insulin and a Subcutaneous Injection of Regular Human Insulin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDC-INS-0002
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Healthy Patients
MeSH Terms: interventions — Insulin

ARMS (4):
- Technosphere insulin inhalation system, 25 units (Experimental)
  Interventions: Drug: Technosphere Insulin
- Technosphere insulin inhalation system, 50 units (Experimental)
  Interventions: Drug: Technosphere insulin
- Technosphere insulin inhalation system, 100 units (Experimental)
  Interventions: Drug: Technosphere insulin
- Subcutaneous regular human insulin (Active Comparator)
  Interventions: Drug: Regular human insulin

INTERVENTIONS:
Drug: Technosphere Insulin
  Arms: Technosphere insulin inhalation system, 25 units
Drug: Technosphere insulin
  Arms: Technosphere insulin inhalation system, 50 units
Drug: Technosphere insulin
  Arms: Technosphere insulin inhalation system, 100 units
Drug: Regular human insulin
  Arms: Subcutaneous regular human insulin

SUMMARY:
A prospective, single center, open randomized, six way crossover study comparing the dose response effect of four different doses of Technosphere Insulin after pulmonary function delivery in comparison to s.c. injection of two different doses of regular human insulin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be in good health, as judge by brief history and physical examination.
* Sex: both, male and female.
* Age: 18-40 years.
* Body mass index: 18-27 kg/m2.
* Capability to reach peak inspiratory flow of >41/sec measured by a computer assisted spirometry.
* FEV1 equal to or greater than 80% of predicted normal.

Exclusion Criteria:

* Diabetes Mellitus type 1 or type 2.
* Human insulin antibodies.
* Anamnestic history of hypersensitivity to the study medication or to drugs with similar chemical structures.
* Having a history of severe or multiple allergies.
* Treatment with any other investigational drug in the last three months before study entry.
* Progressive fatal disease.
* History of significant cardiovascular, respiratory, gastrointestinal, hepatic, renal, neurological, psychiatric and /or hematological disease.
* Having ongoing respiratory tract infection.
* Smoker defined as subjects with evidence or history of tobacco or nicotine use in the last year prior to entry in the study.
* Blood donation within the last 30 days.
* A woman who is lactating.
* Pregnant women or women intending to become pregnant during the study.
* A sexually active woman of childbearing age not actively practicing birth control or using medically accepted device or therapy.
* A lack of compliance or other reasons, which prevent to the opinion of the investigator the participation of the subject in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1999-08; Primary Completion 2000-02 (Actual); Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Dose-corrected area-under-the serum insulin concentration vs. time curve for inhaled TI and subcutaneous RHI at timepoints -120, -90, -60, 0, 1, 3, 7, 12, 20, 30, 45, 60 and 90 minutes, and 2, 3, 4, 5 and 6 hours relative to treatment | crossover every 3-28 days for up to 20 weeks
Area under the glucose infusion rate for inhaled TI and subcutaneous RHI at timepoints -120, -90, -60, 0, 1, 3, 7, 12, 20, 30, 45, 60 and 90 minutes, and 2, 3, 4, 5 and 6 hours relative to treatment | crossover every 3-28 days for up to 20 weeks

SECONDARY OUTCOMES:
Safety variables included adverse events (AEs), clinical laboratory tests, HbA1c, pulmonary function tests, vital signs, physical examinations, and diabetes-specific signs (ie, hypoglycemia) | crossover every 3-28 days for up to 20 weeks